CLINICAL TRIAL: NCT03433781
Title: A Phase Ib Study Evaluating the Safety and Tolerability of Vitamin C in Patients With Intermediate or High Risk Myelodysplastic Syndrome With TET2 Mutations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Perlmutter New York University Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00978
Record Dates: First submitted 2018-02-08; First posted 2018-02-15 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Myelodysplastic Syndromes
Keywords: ASCORBIC ACID
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: 3 dose-escalation cohorts in a 3+3 design. One subject at a time will be enrolled into the first cohort until the first dose level cohort is completed and all patients treated successfully for one cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vitamin C 50 g (Experimental): Patients will receive Vitamin C as a continuous intravenous infusion (CIVI) of 50 grams (g) daily over 24 hours for 5 days for total of 250 grams over 5 days up.
  Interventions: Drug: Vitamin C
- Vitamin C 75 g (Experimental): Patients will receive Vitamin C as a continuous intravenous infusion (CIVI) of 75 grams (g) daily over 24 hours for 5 days for total of 375 grams over 5 days.
  Interventions: Drug: Vitamin C
- Vitamin C 100 g (Experimental): Patients will receive Vitamin C as a continuous intravenous infusion (CIVI) of 100 grams (g) daily over 24 hours for 5 days for total of 500 grams over 5 days.
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Vitamin C — All patients will receive at least 1 cycle of treatment (4 weeks) of Vitamin C as a continuous intravenous infusion (CIVI). Patients with clinical benefit (CR, PR, or SD) then will undergo a second 4-week cycle of treatment. Patients to receive a maximum of 16 weeks of treatment (4 cycles). If a patient progress after receiving a cycle of treatment then the patient will be withdrawn from the study. Patients will be maintained on 1 gram oral Vitamin C daily from the end of the CIVI until the beginning of the next cycle (from day 6 till 28).
  Other Names: ascorbic acid; ascorbate

SUMMARY:
This is an open label, Phase Ib study designed to evaluate the safety, toxicity and biological activity of high dose Vitamin C in bone marrow and peripheral blood when administered as therapy to patients with intermediate or high risk myelodysplastic syndrome according to the revised IPSS (international prognostic scoring system) criteria whose disease has a Ten-eleven translocation-2, (TET2) mutation. The primary objectives phase 1 study is to establish safety and confirm a steady level of Vitamin C on ≥1 mM in > 75% of the patients is achieved. All patients will receive at least 1 cycle of treatment (4 weeks). Patients with clinical benefit (CR,PR, or SD) then will undergo a second 4-week cycle of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed Myelodysplastic Syndrome with positive TET2 mutations (We will test all MDS patients for TET2 mutations using next generation sequencing and only patients with TET2 mutations will be included in our study)
* Myeloblasts account for less than 20% of leukocytes on peripheral blood and bone marrow aspirate
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Appendix 1)
* Adequate organ function

  1. Platelets ≥20,000/μL
  2. Absolute neutrophil count ≥ 500/μL
  3. Bilirubin < 1.5 x institutional upper limit of normal (ULN) or < 3 x ULN in patients with Gilbert's disease or liver involvement
  4. Serum albumin ≥ 2.0 g/dL
  5. Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) ≤2.5 institutional ULN or, in the case of liver involvement by the primary disease AST/ALT ≤ 5 x ULN
  6. Creatinine≤1.5 x institutional ULN or estimated creatinine clearance of ≥45 mL/min by the Cockcroft-Gault equation or measured creatinine clearance >45 mL/min
* Females of child bearing potential must have a negative serum pregnancy test with 7 days prior to first dose of treatment and use 2 methods of contraceptives while on treatment
* Ability to understand and the willingness to sign a written informed consent document
* Patients currently receiving or who previously received Hydroxyurea, Erythrocyte stimulating agents (ESA), or granulocyte colony stimulating factors (G-CSF) are allowed to participate in the study.

Exclusion Criteria:

* Concurrent hypomethylation agent usage; the last dose of treatment must be ≥4 weeks before the start of the Vitamin C infusion
* Myeloblast count ≥20% in peripheral blood or bone marrow aspirate
* Major surgery within 2 weeks prior to first dose of study drug
* Allogeneic stem cell transplant
* Any previous chemotherapy agent other than hypomethylating agents (e.g., Venetoclax)
* Uncontrolled concurrent serious illness
* Concurrent malignancy or history of a previous malignancy within 1 year prior to first dose of the current study, unless curatively resected basal, squamous cell carcinoma of the skin, breast ductal/lobular carcinoma in situ or cervical carcinoma in situ.
* Active infections including hepatitis B carrier status, hepatitis C virus (HCV) infection (patients must have a negative Hep B and Hep C viral load at screening)
* Known HIV-positive status
* Any significant medical conditions, laboratory abnormality, or psychiatric illness that would exclude the subject from participation or interfere with study treatment, monitoring and compliance such as:

  1. Unstable angina pectoris, symptomatic congestive heart failure (NYHA III or IV), myocardial infarction ≤ 6 months prior to first study drug, clinically significant and uncontrolled cardiac arrhythmia (e.g. atrial fibrillation/flutter ventricular cardiovascular physiology is allowed), cerebrovascular accidents ≤ 6 months before study drug start
  2. Severely impaired lung function
* Serious, systemic infection requiring treatment ≤7 days before the first dose of study drug
* Any severe, uncontrolled disease or condition which in the investigator's opinion, may put the subject at significant risk, may confound the study results, or impact the subject's participation in the study
* History of any renal calculi or hyperoxaluria or any other preexisting renal disorder
* History of G6PD deficiency, hereditary spherocytosis or hemochromatosis
* Patients on therapeutic or prophylactic anticoagulation will be excluded from enrollment on the protocol. However, patients can remain on the study if they develop a thrombosis that requires therapeutic anticoagulation during the course of protocol therapy
* Uncontrolled hyponatremia, SIADH, hypokalemia, hyerpkalemia, hypomagnesemia or hypermagnesemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad M Abdul Hay, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - University of Miami Miller School of Medicine -Sylvester Cancer Center, Miami, Florida
  - New York University School of Medicine, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin C 50 g | Vitamin C 75 g | Vitamin C 100 g
Started | 1 | 3 | 0
Completed | 0 | 2 | 0
Not Completed | 1 | 1 | 0
Not completed — Progression of Disease | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled into the Vitamin C 100g arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin C 50 g | Vitamin C 75 g | Vitamin C 100 g | Total
Number analyzed (Participants) | 1 | 3 | 0 | 4
Age, Continuous [Median (Standard Deviation); unit: years] | 73 (0) | 76 (2.49) |  | 74 (2.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 2
  Male | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  | 0
  Not Hispanic or Latino | 1 | 3 |  | 4
  Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 1 |  | 1
  White | 1 | 2 |  | 3
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced a Dose Limiting Toxicity (DLT)
Description: DLT is defined as grade 3 or higher of any duration or as a Grade ≥2 adverse event (AE) that persists for ≥96 hours with the exception of Grade ≥ 2 AEs clearly related to the underlying MDS
Time Frame: Week 16
Population: No patients were enrolled into the Vitamin C 100 g arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin C 50 g | Vitamin C 75 g | Vitamin C 100 g
Number analyzed (Participants) | 1 | 2 | 0
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 years
Description: No patients were enrolled in the Vitamin C 100 g group.
Arm/Group | Vitamin C 50 g | Vitamin C 75 g | Vitamin C 100 g
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin C 50 g (N=1) | Vitamin C 75 g (N=3) | Vitamin C 100 g (N=0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | NA
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA
Catheter Related Infection (Infections and infestations) | 1 (1) | 0 (0) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vitamin C 50 g (N=1) | Vitamin C 75 g (N=3) | Vitamin C 100 g (N=0)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | NA
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT03433781/Prot_SAP_000.pdf